CLINICAL TRIAL: NCT00232180
Title: The Effect Of Eplerenone Versus Placebo On Cardiovascular Mortality And Heart Failure Hospitalization In Subjects With NYHA Class II Chronic Systolic Heart Failure
Brief Title: A Comparison Of Outcomes In Patients In New York Heart Association (NYHA) Class II Heart Failure When Treated With Eplerenone Or Placebo In Addition To Standard Heart Failure Medicines
Acronym: EMPHASIS-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6141079
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure
Keywords: Open-label; single arm mortality/morbidity trial eplerenone chronic systolic heart failure
MeSH Terms: conditions — Heart Failure | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eplerenone arm (Active Comparator): Eplerenone administered on top of background standard heart failure therapy
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — Eplerenone administered on top of background standard heart failure therapy

SUMMARY:
In an earlier study, eplerenone was shown to improve survival in patients who had heart failure immediately following a heart attack. However, it is not known how patients with established mild-to-moderate heart failure (NYHA Class II), who have the additional risk of sudden death, will respond if treated with eplerenone. In this trial, eplerenone plus standard heart failure medicines is being compared to placebo plus standard heart failure medicines in terms of an additional ability to prolong life and prevent re-hospitalizations for worsening heart failure in these patients.

The Data Safety Monitoring Committee (DSMC) observed during its conduct of the protocol-specified second interim analysis on the 6th of May, 2010 that the efficacy of eplerenone had met the pre-specified stopping rules in the protocol. As a result of the discussion between the DSMC and the Executive Steering Committee (ESC), the ESC recommended that EMPHASIS-HF should be terminated, Based on the convincing efficacy and the consideration that it would be unethical not to offer this treatment to patients, the ESC recommended that all the patients in the trial should be transferred to open-label eplerenone. The Open Label Extension eplerenone arm will last for 12 months. Eplerenone is not currently approved for the indication studied in this patient population.

On May 26, 2010, further enrollment into EMPHASIS-HF was stopped. The amendment is considered to be the most appropriate way to ensure that all the subjects who participated in the double-blind phase of the EMPHASIS-HF trial can be offered treatment with eplerenone

ELIGIBILITY:
Inclusion Criteria:

* History (Hx) of chronic systolic heart failure of ischemic or non-ischemic etiology of at least 4 weeks duration; Currently, New York Heart Association (NYHA) functional Class II and on optimal dose, or maximally tolerated dose of standard heart failure medicines (advisable to include ACE-I/ARBs; beta-blockers) and diuretics if indicated for fluid overload. Should have participated in the double-blind phase of the EMPHASIS-HF trial

Exclusion Criteria:

* Severe chronic systolic heart failure symptomatic at rest despite optimal medical therapy; estimated glomerular filtration rate (eGFR) <30 ml/min/1.73m2.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2743 (Actual)
Dates: Start 2006-03; Primary Completion 2010-05 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (247):
- United States (40):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Loma Linda, California
  - Pfizer Investigational Site, Merced, California
  - Pfizer Investigational Site, Stockton, California
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Bridgeport, Connecticut
  - Pfizer Investigational Site, Hartford, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Jupiter, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Bangor, Maine
  - Pfizer Investigational Site, Annapolis, Maryland
  - Pfizer Investigational Site, Columbia, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, MN, Minnesota
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Manchester, New Hampshire
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Beaver, Pennsylvania
  - Pfizer Investigational Site, Doylestown, Pennsylvania
  - Pfizer Investigational Site, Leetsdale, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Cumberland, Rhode Island
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Madison, Wisconsin
- Argentina (3):
  - Pfizer Investigational Site, Morón, Pcia. de Buenos Aires
  - Pfizer Investigational Site, Buenos Aires
  - Pfizer Investigational Site, Córdoba
- Australia (3):
  - Pfizer Investigational Site, Concord, New South Wales
  - Pfizer Investigational Site, Brisbane, Queensland
  - Pfizer Investigational Site, Launceston, Tasmania
- Belgium (11):
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Bonheiden
  - Pfizer Investigational Site, Eupen
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Hasselt
  - Pfizer Investigational Site, Huy
  - Pfizer Investigational Site, La Louvière
  - Pfizer Investigational Site, Lanaken
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Overpelt
  - Pfizer Investigational Site, Yvoir
- Canada (7):
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Saint-Charles-Borromée, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, St-georges (Beauce), Quebec
- Czechia (6):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Ostrava
  - Pfizer Investigational Site, Pilsen
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Příbram
- France (15):
  - Pfizer Investigational Site, Toulouse, Cedex 4
  - Pfizer Investigational Site, Créteil, Cedex
  - Pfizer Investigational Site, Gap, Cedex
  - Pfizer Investigational Site, Angers
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Cergy-Pontoise
  - Pfizer Investigational Site, Châteauroux
  - Pfizer Investigational Site, Gap
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Nîmes
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Saint-Amand-Montrond
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Valenciennes
- Germany (16):
  - Pfizer Investigational Site, Bad Nauheim
  - Pfizer Investigational Site, Bad Rothenfelde
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Dortmund
  - Pfizer Investigational Site, Duisburg
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Frankfurt am Main
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Hagen
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, Homburg/Saar
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Ludwigshafen
  - Pfizer Investigational Site, Lübeck
- Greece (4):
  - Pfizer Investigational Site, Athens, Attica
  - Pfizer Investigational Site, Haidari, Attica
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Thessaloniki
- Hong Kong (3):
  - Pfizer Investigational Site, Chai Wan
  - Pfizer Investigational Site, Pokfulam
  - Pfizer Investigational Site, Shatin NT
- Hungary (5):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Mosonmagyaróvár
  - Pfizer Investigational Site, Siófok
  - Pfizer Investigational Site, Szeged
- India (7):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Pune, Maharshtra
  - Pfizer Investigational Site, Ludhiana, Punjab
  - Pfizer Investigational Site, Chennai, Tamil Nadu
  - Pfizer Investigational Site, Coimbatore, Tamil Nadu
  - Pfizer Investigational Site, Lucknow, Uttar Pradesh
- Ireland (3):
  - Pfizer Investigational Site, Cork
  - Pfizer Investigational Site, Dublin
  - Pfizer Investigational Site, Galway
- Italy (15):
  - Pfizer Investigational Site, Bergamo (BG)
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Mestre - Zelardino (VE)
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Modena
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Parma
  - Pfizer Investigational Site, Piacenza
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Sassari
  - Pfizer Investigational Site, Trieste
  - Pfizer Investigational Site, Venezia
- Mexico (7):
  - Pfizer Investigational Site, Aguascalientes, Aguacalientes
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Zapopan, Jalisco
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Aguascalientes
  - Pfizer Investigational Site, Chihuahua City
  - Pfizer Investigational Site, San Luis Potosí City
- Netherlands (13):
  - Pfizer Investigational Site, 's-Hertogenbosch
  - Pfizer Investigational Site, Alkmaar
  - Pfizer Investigational Site, Apeldoorn
  - Pfizer Investigational Site, Arnhem
  - Pfizer Investigational Site, Breda
  - Pfizer Investigational Site, Deventer
  - Pfizer Investigational Site, Dordrecht
  - Pfizer Investigational Site, Eindhoven
  - Pfizer Investigational Site, Groningen
  - Pfizer Investigational Site, Heerlen
  - Pfizer Investigational Site, Veldhoven
  - Pfizer Investigational Site, Velp
  - Pfizer Investigational Site, Zwolle
- Poland (8):
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Piotrkow Trybunalski
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Stalowa Wola
  - Pfizer Investigational Site, Szczecin
  - Pfizer Investigational Site, Warsaw
- Portugal (11):
  - Pfizer Investigational Site, Guilhufe - PNF, Penafiel
  - Pfizer Investigational Site, Almada
  - Pfizer Investigational Site, Amadora
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Linda a Velha
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Oliveira de Azeméis
  - Pfizer Investigational Site, Portalegre
  - Pfizer Investigational Site, Porto
  - Pfizer Investigational Site, Vila Franca de Xira
  - Pfizer Investigational Site, Vila Real
- Russia (6):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Novosibirsk
  - Pfizer Investigational Site, S-Petersburg
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Voronezh
  - Pfizer Investigational Site, Yaroslavl
- Pfizer Investigational Site, Singapore, Singapore
- Slovakia (5):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Levice
  - Pfizer Investigational Site, Liptovský Mikuláš
  - Pfizer Investigational Site, Nitra
  - Pfizer Investigational Site, Trenčín
- South Africa (6):
  - Pfizer Investigational Site, Soweto, Johannesburg
  - Pfizer Investigational Site, Bloemfontein
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Johannesburg
  - Pfizer Investigational Site, KwaKhangela
  - Pfizer Investigational Site, Kwazulu Natal
- South Korea (3):
  - Pfizer Investigational Site, Republic of Korea, Korea
  - Pfizer Investigational Site, Suwon
  - Pfizer Investigational Site, Taegu
- Spain (6):
  - Pfizer Investigational Site, Santiago de Compostela, LA Coruña
  - Pfizer Investigational Site, Barakaldo, Vizcaya
  - Pfizer Investigational Site, Almería
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Córdoba
  - Pfizer Investigational Site, Málaga
- Sweden (13):
  - Pfizer Investigational Site, Ängelholm
  - Pfizer Investigational Site, Bollnäs
  - Pfizer Investigational Site, Falun
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Halmstad
  - Pfizer Investigational Site, Hässleholm
  - Pfizer Investigational Site, Lindesberg
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Luleå
  - Pfizer Investigational Site, Mölndal
  - Pfizer Investigational Site, Skellefteå
  - Pfizer Investigational Site, Varberg
  - Pfizer Investigational Site, Vaxjo
- Ukraine (10):
  - Pfizer Investigational Site, Simferopol, Autonomous Republic of Crimea
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Donetsk
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kiev
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Lviv
  - Pfizer Investigational Site, Odesa
  - Pfizer Investigational Site, Uzhhorod
  - Pfizer Investigational Site, Zaporizhzhia
- United Arab Emirates (2):
  - Pfizer Investigational Site, Dubai, UAE
  - Pfizer Investigational Site, Abu Dhabi
- United Kingdom (16):
  - Pfizer Investigational Site, Knutsford, Cheshire
  - Pfizer Investigational Site, Macclesfield, Cheshire
  - Pfizer Investigational Site, Belfast, Northern Ireland
  - Pfizer Investigational Site, Glasgow, Strathclyde
  - Pfizer Investigational Site, Belfast
  - Pfizer Investigational Site, Coventry
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Harrow
  - Pfizer Investigational Site, Larbert
  - Pfizer Investigational Site, Macclesfield
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Milton Keynes
  - Pfizer Investigational Site, Sheffield
  - Pfizer Investigational Site, Southend-on-Sea
  - Pfizer Investigational Site, Torquay
- Venezuela (2):
  - Pfizer Investigational Site, Caracas, Distrito Federal
  - Pfizer Investigational Site, Caracas, Miranda

REFERENCES:
- [Derived] Matsumoto S, Kondo T, Jhund PS, Campbell RT, Swedberg K, van Veldhuisen DJ, Pocock SJ, Pitt B, Zannad F, McMurray JJV. Underutilization of Mineralocorticoid Antagonists in Patients With Heart Failure With Reduced Ejection Fraction. J Am Coll Cardiol. 2023 Sep 12;82(11):1080-1091. doi: 10.1016/j.jacc.2023.06.021. PMID 37642608
- [Derived] Vaduganathan M, Ferreira JP, Rossignol P, Neuen BL, Claggett BL, Pfeffer MA, McMurray JJV, Pitt B, Zannad F, Solomon SD. Effects of steroidal mineralocorticoid receptor antagonists on acute and chronic estimated glomerular filtration rate slopes in patients with chronic heart failure. Eur J Heart Fail. 2022 Sep;24(9):1586-1590. doi: 10.1002/ejhf.2635. Epub 2022 Aug 31. PMID 35867859
- [Derived] Martens P, Ferreira JP, Vincent J, Abreu P, Busselen M, Mullens W, Tang WHW, Bohm M, Pitt B, Zannad F, Rossignol P. Prognostic relevance of magnesium alterations in patients with a myocardial infarction and left ventricular dysfunction: insights from the EPHESUS trial. Eur Heart J Acute Cardiovasc Care. 2022 Feb 8;11(2):148-159. doi: 10.1093/ehjacc/zuab111. PMID 35021200
- [Derived] Ferreira JP, Lamiral Z, McMurray JJV, Swedberg K, van Veldhuisen DJ, Vincent J, Rossignol P, Pocock SJ, Pitt B, Zannad F. Impact of Insulin Treatment on the Effect of Eplerenone: Insights From the EMPHASIS-HF Trial. Circ Heart Fail. 2021 Jun;14(6):e008075. doi: 10.1161/CIRCHEARTFAILURE.120.008075. Epub 2021 Jun 15. PMID 34129365
- [Derived] Martens P, Ferreira JP, Vincent J, Abreu P, Busselen M, Mullens W, Tang WWH, Bohm M, Pitt B, Zannad F, Rossignol P. Serum sodium and eplerenone use in patients with a myocardial infarction and left ventricular dysfunction or heart failure: insights from the EPHESUS trial. Clin Res Cardiol. 2022 Apr;111(4):380-392. doi: 10.1007/s00392-021-01853-8. Epub 2021 Apr 23. PMID 33893561
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592
- [Derived] Monzo L, Ferreira JP, Abreu P, Szumski A, Bohm M, McMurray JJV, Pitt B, Swedberg K, van Veldhuisen DJ, Girerd N, Vincent J, Zannad F, Rossignol P. Visit-to-visit blood pressure variation and outcomes in heart failure with reduced ejection fraction: findings from the Eplerenone in Patients with Systolic Heart Failure and Mild Symptoms trial. J Hypertens. 2020 Mar;38(3):420-425. doi: 10.1097/HJH.0000000000002275. PMID 31584516
- [Derived] Stienen S, Ferreira JP, Vincent J, Busselen M, Li B, McMurray JJV, Pitt B, Girerd N, Rossignol P, Zannad F. Estimated Long-Term Survival With Eplerenone. J Am Coll Cardiol. 2019 May 14;73(18):2357-2359. doi: 10.1016/j.jacc.2019.02.043. No abstract available. PMID 31072582
- [Derived] Ferreira JP, Duarte K, McMurray JJV, Pitt B, van Veldhuisen DJ, Vincent J, Ahmad T, Tromp J, Rossignol P, Zannad F. Data-Driven Approach to Identify Subgroups of Heart Failure With Reduced Ejection Fraction Patients With Different Prognoses and Aldosterone Antagonist Response Patterns. Circ Heart Fail. 2018 Jul;11(7):e004926. doi: 10.1161/CIRCHEARTFAILURE.118.004926. PMID 29997240
- [Derived] Rossignol P, Dobre D, McMurray JJ, Swedberg K, Krum H, van Veldhuisen DJ, Shi H, Messig M, Vincent J, Girerd N, Bakris G, Pitt B, Zannad F. Incidence, determinants, and prognostic significance of hyperkalemia and worsening renal function in patients with heart failure receiving the mineralocorticoid receptor antagonist eplerenone or placebo in addition to optimal medical therapy: results from the Eplerenone in Mild Patients Hospitalization and Survival Study in Heart Failure (EMPHASIS-HF). Circ Heart Fail. 2014 Jan;7(1):51-8. doi: 10.1161/CIRCHEARTFAILURE.113.000792. Epub 2013 Dec 2. PMID 24297687
- [Derived] Eschalier R, McMurray JJ, Swedberg K, van Veldhuisen DJ, Krum H, Pocock SJ, Shi H, Vincent J, Rossignol P, Zannad F, Pitt B; EMPHASIS-HF Investigators. Safety and efficacy of eplerenone in patients at high risk for hyperkalemia and/or worsening renal function: analyses of the EMPHASIS-HF study subgroups (Eplerenone in Mild Patients Hospitalization And SurvIval Study in Heart Failure). J Am Coll Cardiol. 2013 Oct 22;62(17):1585-93. doi: 10.1016/j.jacc.2013.04.086. Epub 2013 Jun 27. PMID 23810881
- [Derived] Krum H, Shi H, Pitt B, McMurray J, Swedberg K, van Veldhuisen DJ, Vincent J, Pocock S, Zannad F; EMPHASIS-HF Study Group. Clinical benefit of eplerenone in patients with mild symptoms of systolic heart failure already receiving optimal best practice background drug therapy: analysis of the EMPHASIS-HF study. Circ Heart Fail. 2013 Jul;6(4):711-8. doi: 10.1161/CIRCHEARTFAILURE.112.000173. Epub 2013 Apr 26. PMID 23625945
- [Derived] Rogers JK, McMurray JJ, Pocock SJ, Zannad F, Krum H, van Veldhuisen DJ, Swedberg K, Shi H, Vincent J, Pitt B. Eplerenone in patients with systolic heart failure and mild symptoms: analysis of repeat hospitalizations. Circulation. 2012 Nov 6;126(19):2317-23. doi: 10.1161/CIRCULATIONAHA.112.110536. Epub 2012 Oct 5. PMID 23042980
- [Derived] Zannad F, McMurray JJ, Krum H, van Veldhuisen DJ, Swedberg K, Shi H, Vincent J, Pocock SJ, Pitt B; EMPHASIS-HF Study Group. Eplerenone in patients with systolic heart failure and mild symptoms. N Engl J Med. 2011 Jan 6;364(1):11-21. doi: 10.1056/NEJMoa1009492. Epub 2010 Nov 14. PMID 21073363
- [Derived] Zannad F, McMurray JJ, Drexler H, Krum H, van Veldhuisen DJ, Swedberg K, Shi H, Vincent J, Pitt B. Rationale and design of the Eplerenone in Mild Patients Hospitalization And SurvIval Study in Heart Failure (EMPHASIS-HF). Eur J Heart Fail. 2010 Jun;12(6):617-22. doi: 10.1093/eurjhf/hfq049. Epub 2010 Apr 13. PMID 20388647
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6141079&StudyName=The%20Effect%20Of%20Eplerenone%20Versus%20Placebo%20On%20Cardiovascular%20Mortality%20And%20Heart%20Failure%20Hospitalization%20In%20Subjects%20With%20NYHA%20Class%20II%20Chronic%20Systolic%20Heart%20Failure

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1597 participants who completed the double-blind phase, 1246 entered into the open-label phase and 351 participants were ineligible to participate the open-label phase.
Groups:
- Eplerenone: Double-blind Phase: Eplerenone 25 milligram (mg) tablet orally once daily on top of standard heart failure therapy. Dose might have been increased at Week 4 to 50 mg once daily. For participants with an estimated glomerular filtration rate (eGFR) between 30 to 49 milliliter per minute divided by 1.73 squared meter (ml/min/1.73m^2), initial dose was 25 mg orally once every other day; at Week 4, dose might have been increased to a maximum of 25 mg once daily based on serum potassium level.
- Placebo: Double-blind Phase: Placebo matching to eplerenone 25 mg orally once daily on top of standard heart failure therapy.
- Eplerenone: Open Label Phase: Participants from double blind phase received eplerenone 25 mg tablet orally once daily on top of standard heart failure therapy for 12 months. Dose might have been increased at Week 4 to 50 mg once daily. For participants with an eGFR between 30 to 49 ml/min/1.73m^2 in the double blind phase, initial dose was 25 mg orally once every other day; at Week 4, dose might had been increased to a maximum of 25 mg once daily based on serum potassium level.
Period: Double-blind (DB) Phase
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase | Eplerenone: Open Label Phase
Started | 1367 (Three participants in each arm were enrolled after data cut-off.) | 1376 (Three participants in each arm were enrolled after data cut-off.) | 0
Treated | 1364 | 1372 | 0
Completed | 826 | 771 | 0
Not Completed | 541 | 605 | 0
Not completed — Death | 186 | 222 | 0
Not completed — Lost to Follow-up | 34 | 28 | 0
Not completed — Withdrawal by Subject | 131 | 148 | 0
Not completed — Protocol Violation | 28 | 21 | 0
Not completed — Adverse Event | 83 | 100 | 0
Not completed — Other | 70 | 75 | 0
Not completed — Randomized but not treated | 3 | 4 | 0
Not completed — Laboratory abnormality | 6 | 7 | 0
Period: Open Label Phase
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase | Eplerenone: Open Label Phase
Started | 0 | 0 | 1246
Treated | 0 | 0 | 1245
Completed | 0 | 0 | 1098
Not Completed | 0 | 0 | 148
Not completed — Death | 0 | 0 | 48
Not completed — Lost to Follow-up | 0 | 0 | 5
Not completed — Protocol Violation | 0 | 0 | 3
Not completed — Study terminated by sponsor | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 37
Not completed — Other | 0 | 0 | 16
Not completed — Adverse Event | 0 | 0 | 25
Not completed — Laboratory abnormality | 0 | 0 | 10
Not completed — Randomized but not treated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Eplerenone: Eplerenone 25 milligram (mg) tablet orally once daily on top of standard heart failure therapy. Dose might have been increased at Week 4 to 50 mg once daily. For participants with an estimated glomerular filtration rate (eGFR) between 30 to 49 milliliter per minute divided by 1.73 squared meter (ml/min/1.73m^2), initial dose was 25 mg orally once every other day; at Week 4, dose might have been increased to a maximum of 25 mg once daily based on serum potassium level.
- Placebo: Placebo matching to eplerenone 25 mg orally once daily on top of standard heart failure therapy.
- Total: Total of all reporting groups
Arm/Group | Eplerenone | Placebo | Total
Number analyzed (Participants) | 1367 | 1376 | 2743
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 443 | 441 | 884
  65 to 74 years | 594 | 607 | 1201
  75 to 84 years | 302 | 299 | 601
  Greater than or equal to (>=) 85 years | 28 | 29 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 309 | 302 | 611
  Male | 1058 | 1074 | 2132

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of Cardiovascular (CV) Mortality or Hospitalization Due to Heart Failure (HF) (Adjudicated): Up to Cut-off Date
Description: CV mortality is defined as death due to heart failure, myocardial infarction, cardiac arrhythmia, stroke or cerebral vascular accident (CVA), other CV cause (such as aneurysm or pulmonary embolism). Hospitalization due to HF is defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility) due to HF as the primary reason for hospitalization as determined by the endpoint committee adjudicator.
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010)
Population: Full analysis set (FAS) using intent-to-treat (ITT) principle: All randomized participants, followed for mortality, other major endpoints for duration of double blind treatment period, regardless of compliance with study drug and protocol. Here 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1364 | 1373
participants | 249 | 356
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; Cox proportional hazard model includes treatment as the major factor, adjusting for age, estimated glomerular filtration rate, left ventricular ejection fraction, body mass index, hemoglobin, heart rate, systolic blood pressure, diabetes, history of hypertension, prior myocardial infarction, baseline left bundle branch block, time from electrocardiogram Q wave to the end of the S wave corresponding to ventricle depolarization (QRS) and atrial fibrillation as covariates; Test type: Superiority or Other; p < 0.0001, Cox proportional hazard model — Using an adaptation of Haybittle-Peto stopping criterion adjusting for two interim analyses, p-value for final primary analysis will be compared to alpha=0.049. No adjustment in alpha will be made on parameters/endpoints other than primary endpoint; Hazard Ratio (HR) = 0.630, 95% CI 2-sided [0.535 to 0.741]

2. Primary Outcome: Number of Participants With First Occurrence of Cardiovascular (CV) Mortality or Hospitalization Due to Heart Failure (HF) (Adjudicated)
Description: as for outcome 1
Time Frame: Baseline (30 March 2006) up to 59.5 months (complete DB phase: 18 March 2011)
Population: FAS using ITT principle: All randomized participants, followed for mortality and other major endpoints for the duration of the double blind treatment period, regardless of compliance with the study drug and the protocol.
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants | 288 | 392

3. Secondary Outcome: Number of Participants With First Occurrence of All-Cause Mortality or Heart Failure (HF) Hospitalization (Adjudicated)
Description: Death due to any cause or first of occurrence HF hospitalization. HF hospitalization is defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility) due to HF as the primary reason for hospitalization as determined by the endpoint committee adjudicator.
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: FAS using ITT principle: All randomized participants, followed for mortality and other major endpoints for the duration of the double blind treatment period, regardless of compliance with the study drug and the protocol. Here "n" signifies participants evaluated at that time point.
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants
  Up to 50 months (cut-off) (n= 1364, 1373) | 270 | 376
  Up to 59.5 months (complete DB) (n= 1367, 1376) | 311 | 418
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; The statistical analysis was only performed on the adjudicated endpoint data up to cut-off. Cox proportional hazard model includes treatment as the major factor, adjusting for age, estimated glomerular filtration rate, left ventricular ejection fraction, body mass index, hemoglobin, heart rate, systolic blood pressure, diabetes, history of hypertension, prior myocardial infarction, baseline left bundle branch block, QRS complex and atrial fibrillation as covariates; Test type: Superiority or Other; p < 0.0001, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 0.647, 95% CI 2-sided [0.552 to 0.757]

4. Secondary Outcome: Number of Participants With First Occurrence of All-Cause Mortality (Adjudicated)
Description: Death due to any cause.
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants
  Up to 50 months (cut-off) (n= 1364, 1373) | 171 | 213
  Up to 59.5 months (complete DB) (n= 1367, 1376) | 205 | 253
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0081, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 0.761, 95% CI 2-sided [0.622 to 0.932]

5. Secondary Outcome: Number of Participants With First Occurrence of Cardiovascular (CV) Mortality (Adjudicated)
Description: CV mortality is defined as death due to heart failure, myocardial infarction, cardiac arrhythmia, stroke or cerebral vascular accident (CVA), other CV cause (such as aneurysm or pulmonary embolism).
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants
  Up to 50 months (cut-off) (n= 1364, 1373) | 147 | 185
  Up to 59.5 months (complete DB) (n= 1367, 1376) | 178 | 215
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0120, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 0.757, 95% CI 2-sided [0.609 to 0.941]

6. Secondary Outcome: Number of Participants With First Occurrence of All-Cause Hospitalization (Adjudicated)
Description: Hospitalization due to any cause is defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility).
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants
  Up to 50 months (cut-off) (n= 1364, 1373) | 408 | 491
  Up to 59.5 months (complete DB) (n= 1367, 1376) | 463 | 552
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 0.768, 95% CI 2-sided [0.673 to 0.876]

7. Secondary Outcome: Number of Participants With First Occurrence of Heart Failure (HF) Hospitalization (Adjudicated)
Description: First occurrence of HF hospitalization. Hospitalization due to HF is defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility) due to HF as the primary reason for hospitalization as determined by the endpoint committee adjudicator.
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants
  Up to 50 months (cut-off) (n= 1364, 1373) | 164 | 253
  Up to 59.5 months (complete DB) (n= 1367, 1376) | 186 | 277
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 0.576, 95% CI 2-sided [0.473 to 0.702]

8. Secondary Outcome: Number of Participants With First Occurrence of All-Cause Mortality or All-Cause Hospitalization (Adjudicated)
Description: Death due to any cause or hospitalization due to any cause. Hospitalization due to any cause is defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility).
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants
  Up to 50 months (cut-off) (n= 1364, 1373) | 462 | 569
  Up to 59.5 months (complete DB) (n= 1367, 1376) | 530 | 636
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 0.751, 95% CI 2-sided [0.664 to 0.849]

9. Secondary Outcome: Number of Participants With First Occurrence Of Heart Failure (HF) Mortality or Heart Failure (HF) Hospitalization (Adjudicated)
Description: Death due to HF or first occurrence of HF hospitalization. Hospitalization due to HF is defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility) due to HF as the primary reason for hospitalization as determined by the endpoint committee adjudicator.
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants
  Up to 50 months (cut-off) (n= 1364, 1373) | 170 | 262
  Up to 59.5 months (complete DB) (n= 1367, 1376) | 194 | 287
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 0.577, 95% CI 2-sided [0.475 to 0.701]

10. Secondary Outcome: Number of Participants With First Occurrence of Cardiovascular (CV) Hospitalization (Adjudicated)
Description: First occurrence of CV hospitalization. CV hospitalization is defined as hospitalization due to HF (first or subsequent), acute myocardial infarction, angina pectoris (unstable), cardiac arrhythmia (atrial fibrillation [AF], atrial flutter, supraventricular arrhythmias, or ventricular arrhythmias), stroke/CVA, other CV reasons (such as hypotension or peripheral vascular disease), implantation of a cardioverter defibrillator (ICD), or cardiac resynchronization therapy (CRT) with CV event as the primary reason for hospitalization as determined by endpoint committee adjudicator.
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants
  Up to 50 months (cut-off) (n= 1364, 1373) | 304 | 399
  Up to 59.5 months (complete DB) (n= 1367, 1376) | 346 | 439
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 0.694, 95% CI 2-sided [0.598 to 0.806]

11. Secondary Outcome: Number of Participants With First Occurrence of Fatal or Non-fatal Myocardial Infarction (Adjudicated)
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants
  Up to 50 months (cut-off) (n= 1364, 1373) | 45 | 33
  Up to 59.5 months (complete DB) (n= 1367, 1376) | 49 | 40
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2321, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 1.316, 95% CI 2-sided [0.839 to 2.064]

12. Secondary Outcome: Number of Participants With First Occurrence of Fatal or Non-fatal Stroke (Adjudicated)
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants
  Up to 50 months (cut-off) (n= 1364, 1373) | 21 | 26
  Up to 59.5 months (complete DB) (n= 1367, 1376) | 24 | 31
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.4213, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 0.789, 95% CI 2-sided [0.443 to 1.406]

13. Secondary Outcome: Number of Participants With First Occurrence of Implantation of Cardiac Defibrillator (ICD) (Adjudicated)
Description: First occurrence of implantation of cardiac defibrillator (ICD). ICD is an electronic device capable of monitoring the heart rhythm. When the heart is beating normally, the device remains inactive. If the heart develops a life-threatening tachycardia, the ICD delivers electrical shocks to the heart to terminate the abnormal rhythm and return the heart rhythm to normal.
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants
  Up to 50 months (cut-off) (n= 1364, 1373) | 61 | 59
  Up to 59.5 months (complete DB) (n= 1367, 1376) | 76 | 78
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.9754, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 0.994, 95% CI 2-sided [0.694 to 1.424]

14. Secondary Outcome: Number of Participants With First Occurrence of Implantation of Resynchronization Device (Cardiac Resynchronization Therapy [CRT]) (Adjudicated)
Description: First occurrence of implantation of resynchronization device. CRT is use of a specialized pacemaker to re-coordinate the action of the right and left ventricles in heart failure.
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants
  Up to 50 months (cut-off) (n= 1364, 1373) | 33 | 41
  Up to 59.5 months (complete DB) (n= 1367, 1376) | 45 | 53
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2652, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 0.770, 95% CI 2-sided [0.485 to 1.220]

15. Secondary Outcome: Number of Participants With First Occurrence of Hospitalization Due to Worsening Renal Function (Adjudicated)
Description: First occurrence of hospitalization due to worsening renal function. Hospitalization due to worsening renal function is defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility) due to worsening renal function as the primary reason for hospitalization as determined by endpoint committee adjudicator. Worsening renal function is defined as doubling of serum creatinine level from baseline level.
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants
  Up to 50 months (cut-off) (n= 1364, 1373) | 9 | 8
  Up to 59.5 months (complete DB) (n= 1367, 1376) | 10 | 10
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.9537, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 0.971, 95% CI 2-sided [0.366 to 2.578]

16. Secondary Outcome: Number of Participants With First Occurrence of Hospitalization Due to Hyperkalemia (Adjudicated)
Description: First occurrence of hospitalization due to hyperkalemia. Hospitalization due to hyperkalemia is defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility) due to hyperkalemia as the primary reason for hospitalization as determined by endpoint committee adjudicator. Hyperkalemia is defined as serum potassium level greater than (>) 5.5 milliequivalents per liter (mEq/L).
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 1367 | 1376
participants
  Up to 50 months (cut-off) (n= 1364, 1373) | 4 | 3
  Up to 59.5 months (complete DB) (n= 1367, 1376) | 4 | 3
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8539, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 1.154, 95% CI 2-sided [0.251 to 5.312]

17. Secondary Outcome: Number of Participants With New Onset Atrial Fibrillation or Flutter
Description: New onset of atrial fibrillation or flutter is defined as the diagnosis of atrial fibrillation or flutter in a participant after randomization, where atrial fibrillation was not present before randomization.
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: FAS using ITT principle: Here 'N' (Number of Participants Analyzed) signifies those who did not report a history of atrial fibrillation at baseline and "n" signifies participants evaluated at that time point.
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 956 | 940
participants
  Up to 50 months (cut-off) (n= 950, 937) | 32 | 52
  Up to 59.5 months (complete DB) (n= 956, 940) | 41 | 59
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0175, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 0.585, 95% CI 2-sided [0.376 to 0.910]

18. Secondary Outcome: Number of Participants With New Onset Diabetes Mellitus (DM)
Description: The definition of new onset diabetes mellitus is the diagnosis of diabetes mellitus in a participant after randomization, when DM was not present before randomization.
Time Frame: Baseline (30 March 2006) up to 50 months (cut-off date: 25 May 2010), 59.5 months (complete DB phase: 18 March 2011)
Population: FAS using ITT principle: Here 'N' (Number of Participants Analyzed) signifies those who did not report a history of diabetes mellitus at baseline and "n" signifies participants evaluated at that time point.
Measure: Number; unit: participants
Arm/Group | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase
Number analyzed (Participants) | 907 | 975
participants
  Up to 50 months (cut-off) (n= 904, 973) | 34 | 40
  Up to 59.5 months (complete DB) (n= 907, 975) | 42 | 47
Statistical Analysis 1: Comparison: Eplerenone: Double-blind Phase vs Placebo: Double-blind Phase; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.6009, Cox proportional hazard model — Statistically significant if p-value <0.01; Hazard Ratio (HR) = 0.885, 95% CI 2-sided [0.559 to 1.400]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. The numbers of subjects with each AE or SAE are summarized. If a subject had multiple episodes of the same AE or SAE during the study, only the most severe case of the AE or SAE for the subject are summarized.
Groups:
- Eplerenone: Double-blind Phase (May 25, 2010 Data Cut-off): Eplerenone 25 milligram (mg) tablet orally once daily on top of standard heart failure therapy. Dose might have been increased at Week 4 to 50 mg once daily. For participants with an estimated glomerular filtration rate (eGFR) between 30 to 49 milliliter per minute divided by 1.73 squared meter (ml/min/1.73m^2), initial dose was 25 mg orally once every other day; at Week 4, dose might have been increased to a maximum of 25 mg once daily based on serum potassium level.
- Placebo: Double-blind Phase(May 25, 2010 Data Cutoff); Placebo: Double-blind Phase: Placebo matching to eplerenone 25 mg orally once daily on top of standard heart failure therapy.
- Eplerenone: Double-blind Phase: Eplerenone 25 milligram (mg) tablet orally once daily on top of standard heartfailure therapy. Dose might have been increased at Week 4 to 50 mg once daily.For participants with an estimated glomerular filtration rate (eGFR) between 30 to49 milliliter per minute divided by 1.73 squared meter (ml/min/1.73m^2), initialdose was 25 mg orally once every other day; at Week 4, dose might have beenincreased to a maximum of 25 mg once daily based on serum potassium level.
Arm/Group | Eplerenone: Double-blind Phase (May 25, 2010 Data Cut-off) | Placebo: Double-blind Phase(May 25, 2010 Data Cutoff) | Eplerenone: Double-blind Phase | Placebo: Double-blind Phase | Eplerenone: Open Label Phase
Serious Adverse Events (participants affected / at risk) | 509/1360 | 614/1369 | 586/1364 | 686/1372 | 251/1245
Other Adverse Events (participants affected / at risk) | 547/1360 | 540/1369 | 640/1364 | 617/1372 | 329/1245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eplerenone: Double-blind Phase (May 25, 2010 Data Cut-off) (N=1360) | Placebo: Double-blind Phase(May 25, 2010 Data Cutoff) (N=1369) | Eplerenone: Double-blind Phase (N=1364) | Placebo: Double-blind Phase (N=1372) | Eplerenone: Open Label Phase (N=1245)
Anaemia (Blood and lymphatic system disorders) | 10 | 7 | 12 | 9 | 6
Coagulopathy (Blood and lymphatic system disorders) | 1 | 3 | 1 | 3 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 3 | 2 | 5 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 3 | 0 | 3 | 0
Acute myocardial infarction (Cardiac disorders) | 11 | 8 | 11 | 10 | 11
Angina pectoris (Cardiac disorders) | 9 | 13 | 11 | 18 | 5
Angina unstable (Cardiac disorders) | 24 | 23 | 27 | 30 | 9
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 9 | 20 | 10 | 20 | 2
Arrhythmia supraventricular (Cardiac disorders) | 2 | 0 | 2 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 22 | 30 | 28 | 33 | 7
Atrial flutter (Cardiac disorders) | 5 | 7 | 5 | 7 | 5
Atrial tachycardia (Cardiac disorders) | 0 | 2 | 0 | 3 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 2 | 6 | 3 | 6 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 2 | 0 | 2 | 0
Bradyarrhythmia (Cardiac disorders) | 2 | 3 | 3 | 3 | 0
Bradycardia (Cardiac disorders) | 5 | 4 | 5 | 4 | 3
Bundle branch block left (Cardiac disorders) | 2 | 1 | 2 | 1 | 0
Cardiac aneurysm (Cardiac disorders) | 0 | 1 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 13 | 15 | 15 | 17 | 2
Cardiac asthma (Cardiac disorders) | 3 | 2 | 3 | 2 | 0
Cardiac failure (Cardiac disorders) | 187 | 243 | 218 | 270 | 44
Cardiac failure acute (Cardiac disorders) | 1 | 3 | 1 | 5 | 3
Cardiac failure chronic (Cardiac disorders) | 2 | 4 | 2 | 4 | 1
Cardiac failure congestive (Cardiac disorders) | 13 | 19 | 14 | 18 | 6
Cardiac perforation (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 1 | 1 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 4 | 2
Cardiogenic shock (Cardiac disorders) | 4 | 6 | 5 | 6 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 2 | 0 | 2 | 1
Cardiopulmonary failure (Cardiac disorders) | 3 | 3 | 3 | 3 | 0
Cardiovascular disorder (Cardiac disorders) | 2 | 1 | 3 | 1 | 0
Conduction disorder (Cardiac disorders) | 2 | 3 | 3 | 3 | 0
Congestive cardiomyopathy (Cardiac disorders) | 3 | 1 | 3 | 1 | 0
Coronary artery disease (Cardiac disorders) | 6 | 4 | 7 | 5 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 5 | 1 | 6 | 4 | 1
Coronary artery thrombosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 2 | 2 | 2 | 2 | 3
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 1 | 2
Left ventricular failure (Cardiac disorders) | 6 | 6 | 5 | 10 | 1
Low cardiac output syndrome (Cardiac disorders) | 1 | 0 | 1 | 1 | 0
Mitral valve disease (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 29 | 29 | 36 | 34 | 6
Myocardial ischaemia (Cardiac disorders) | 5 | 3 | 5 | 3 | 1
Palpitations (Cardiac disorders) | 1 | 3 | 1 | 3 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 1 | 1 | 0
Pericardial haemorrhage (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 3 | 1 | 3 | 0
Sinus arrest (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 1 | 3 | 1 | 0
Tachycardia (Cardiac disorders) | 5 | 4 | 5 | 4 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 3 | 2 | 4 | 3 | 3
Ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 10 | 8 | 11 | 10 | 4
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 17 | 27 | 19 | 33 | 8
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 1 | 1 | 0
Haematotympanum (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 1 | 0 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 2 | 1 | 2 | 2 | 2
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1 | 0 | 0
Amaurosis fugax (Eye disorders) | 1 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 2 | 1 | 3 | 0
Diplopia (Eye disorders) | 1 | 0 | 1 | 0 | 0
Phacolytic glaucoma (Eye disorders) | 0 | 1 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 1 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 0 | 0 | 1
Thyroid disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 5 | 2 | 6 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 2 | 3 | 2 | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 2
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 4 | 2 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1 | 2 | 2 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 3 | 4 | 4 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 4 | 3 | 4 | 3 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Pancreatolithiasis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Proctitis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3 | 2 | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mesenteric occlusion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pancreatic insufficiency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 6 | 2 | 6 | 1
Cardiac death (General disorders) | 0 | 2 | 0 | 2 | 0
Chest pain (General disorders) | 21 | 28 | 22 | 31 | 7
Condition aggravated (General disorders) | 0 | 1 | 0 | 2 | 0
Crepitations (General disorders) | 0 | 1 | 0 | 1 | 0
Death (General disorders) | 26 | 34 | 39 | 50 | 12
Device breakage (General disorders) | 0 | 0 | 1 | 0 | 1
Device dislocation (General disorders) | 0 | 1 | 0 | 1 | 0
Device lead damage (General disorders) | 1 | 0 | 1 | 0 | 0
Device malfunction (General disorders) | 2 | 1 | 2 | 1 | 2
Device occlusion (General disorders) | 1 | 1 | 1 | 1 | 0
Device pacing issue (General disorders) | 0 | 1 | 0 | 1 | 0
Device stimulation issue (General disorders) | 0 | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 1
General physical health deterioration (General disorders) | 5 | 2 | 5 | 3 | 0
Hyperplasia (General disorders) | 0 | 0 | 0 | 1 | 1
Impaired healing (General disorders) | 1 | 0 | 1 | 0 | 1
Implant site discharge (General disorders) | 0 | 0 | 0 | 1 | 0
Lipogranuloma (General disorders) | 1 | 0 | 1 | 0 | 0
Malaise (General disorders) | 2 | 1 | 2 | 1 | 0
Mass (General disorders) | 0 | 1 | 0 | 1 | 0
Medical device complication (General disorders) | 0 | 1 | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 2 | 1 | 3 | 0
Necrosis (General disorders) | 1 | 0 | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 3 | 1 | 3 | 1
Pain (General disorders) | 1 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 5 | 1 | 4 | 0
Spinal pain (General disorders) | 0 | 0 | 0 | 1 | 0
Sudden cardiac death (General disorders) | 5 | 11 | 8 | 12 | 4
Sudden death (General disorders) | 10 | 24 | 15 | 24 | 7
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 2 | 0 | 2 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 2 | 0 | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 4 | 1 | 4 | 3 | 2
Cholecystitis acute (Hepatobiliary disorders) | 2 | 3 | 2 | 3 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 5 | 2 | 5 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 1 | 1 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 1
Hepatorenal failure (Hepatobiliary disorders) | 2 | 0 | 2 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 2 | 0 | 3 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 1 | 1 | 1 | 1 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Breast abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 6 | 12 | 6 | 13 | 2
Bronchopneumonia (Infections and infestations) | 4 | 4 | 6 | 5 | 1
Cellulitis (Infections and infestations) | 3 | 2 | 4 | 2 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 1 | 1 | 2 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Dermo-hypodermitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 3 | 1 | 1 | 2 | 2
Diabetic gangrene (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 1 | 1 | 1
Endocarditis (Infections and infestations) | 0 | 2 | 0 | 2 | 1
Erysipelas (Infections and infestations) | 0 | 6 | 0 | 7 | 0
Gangrene (Infections and infestations) | 3 | 0 | 4 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 3 | 6 | 3 | 4
Haematoma infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hepatobiliary infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Implant site infection (Infections and infestations) | 0 | 1 | 2 | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 2 | 1 | 4 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 2 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 1 | 1 | 1 | 0
Joint tuberculosis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 1 | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 4 | 4 | 5 | 2
Lung infection (Infections and infestations) | 2 | 1 | 2 | 2 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Orchitis (Infections and infestations) | 1 | 1 | 1 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Phlebitis infective (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 22 | 29 | 29 | 32 | 17
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 1 | 2 | 1 | 0
Respiratory tract infection (Infections and infestations) | 3 | 8 | 3 | 12 | 2
Sepsis (Infections and infestations) | 3 | 3 | 3 | 4 | 2
Septic shock (Infections and infestations) | 7 | 6 | 7 | 7 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 2 | 0 | 2 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1 | 1 | 2 | 0
Systemic candida (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 3
Urinary tract infection (Infections and infestations) | 7 | 6 | 8 | 10 | 3
Urosepsis (Infections and infestations) | 3 | 2 | 3 | 4 | 1
Viral infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Wound infection (Infections and infestations) | 0 | 2 | 0 | 2 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes zoster ophthalmic (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Joint abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tuberculous laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infected sebaceous cyst (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 8 | 10 | 9 | 12 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 2 | 3 | 4 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2 | 0
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1
Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0 | 2
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 2 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 0 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Arteriogram (Investigations) | 1 | 0 | 1 | 0 | 0
Arteriogram coronary (Investigations) | 1 | 3 | 1 | 3 | 0
Arthroscopy (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 2 | 1 | 2 | 0
Blood glucose abnormal (Investigations) | 1 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 1 | 0
Blood urea increased (Investigations) | 1 | 0 | 1 | 1 | 0
Carotid bruit (Investigations) | 1 | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 1 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0
International normalised ratio decreased (Investigations) | 0 | 1 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 2 | 1 | 3 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 1 | 1 | 1
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 3 | 8 | 3 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 2 | 6 | 2 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 0
Gout (Metabolism and nutrition disorders) | 5 | 2 | 6 | 2 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 2 | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 16 | 7 | 19 | 7 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 4 | 3 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 5 | 4 | 6 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 2 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1 | 4 | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Podagra (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 3 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 2 | 7 | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 2 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1 | 2 | 0
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 2 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2 | 2 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 3 | 0 | 0
Bronchial neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 2 | 4 | 2
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 4 | 1 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 3
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 4 | 2 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4 | 4 | 4 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 2 | 0
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 1 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 4 | 4 | 4
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Pleura carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Brain injury (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Carotid artery disease (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 3 | 1 | 3 | 1 | 1
Cerebral atrophy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1 | 1 | 2 | 0
Cerebral infarction (Nervous system disorders) | 1 | 2 | 2 | 2 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 1 | 1 | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 15 | 19 | 20 | 22 | 4
Coma (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 2 | 1 | 2 | 0
Dementia (Nervous system disorders) | 1 | 1 | 1 | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 6 | 3 | 5 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Epilepsy (Nervous system disorders) | 2 | 0 | 2 | 0 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Hemianopia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Ischaemic stroke (Nervous system disorders) | 3 | 6 | 3 | 7 | 4
Loss of consciousness (Nervous system disorders) | 1 | 2 | 3 | 3 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Parkinsonism (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 3 | 0 | 4 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Spinal cord disorder (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Spinal cord ischaemia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 25 | 21 | 26 | 22 | 6
Transient ischaemic attack (Nervous system disorders) | 7 | 9 | 7 | 9 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 2 | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 2 | 3 | 3 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
Depression (Psychiatric disorders) | 1 | 2 | 2 | 2 | 1
Drug dependence (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Pseudodementia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Somatoform disorder cardiovascular (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Panic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Cardiac neurosis (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0
Bladder mass (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 2 | 2 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Pyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 7 | 13 | 10 | 17 | 3
Renal failure acute (Renal and urinary disorders) | 7 | 8 | 9 | 10 | 3
Renal failure chronic (Renal and urinary disorders) | 2 | 0 | 2 | 1 | 0
Renal impairment (Renal and urinary disorders) | 25 | 18 | 27 | 21 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 2
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 8 | 8 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Brain hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cheyne-Stokes respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 7 | 8 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 28 | 16 | 29 | 3
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 4 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 2 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 2 | 0
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 5 | 7 | 2
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 5 | 6 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 11 | 7 | 12 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 2 | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 1
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 2
Aortic aneurysm repair (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
Bladder operation (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
Cardiac ablation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 2 | 1 | 5 | 1
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 1
Cardiac pacemaker revision (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 | 5 | 1 | 6 | 0
Cardiovascular event prophylaxis (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
Cardioversion (Surgical and medical procedures) | 2 | 1 | 2 | 1 | 0
Cataract operation (Surgical and medical procedures) | 0 | 1 | 1 | 1 | 0
Cervical conisation (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Colectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Coronary angioplasty (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
Coronary artery bypass (Surgical and medical procedures) | 0 | 3 | 0 | 3 | 1
Foot amputation (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
Gallbladder operation (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
Heart transplan (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 2 | 0 | 2 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 8 | 12 | 10 | 13 | 0
Inguinal hernia repair (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Lipoma excision (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
Lung lobectomy (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Lung neoplasm surgery (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
Medical device implantation (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Mitral valve repair (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
Mitral valve replacement (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
Prophylaxis (Surgical and medical procedures) | 3 | 1 | 3 | 1 | 0
Renal transplant (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Therapeutic procedure (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Thrombolysis (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
Vascular operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Aortic valve replacement (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Hip surgery (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Implantable defibrillator replacement (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 3 | 3 | 4 | 2 | 2
Aortic aneurysm rupture (Vascular disorders) | 1 | 0 | 1 | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 2 | 0 | 2 | 0
Arterial disorder (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Arterial insufficiency (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Arteritis (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 4 | 2 | 4 | 4 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Embolism (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Extremity necrosis (Vascular disorders) | 3 | 0 | 3 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 1 | 1 | 1 | 1
Haematoma (Vascular disorders) | 2 | 3 | 3 | 3 | 1
Hypertension (Vascular disorders) | 5 | 3 | 5 | 6 | 1
Hypertensive crisis (Vascular disorders) | 1 | 3 | 1 | 5 | 1
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 3 | 6 | 2 | 10 | 3
Iliac artery occlusion (Vascular disorders) | 1 | 1 | 2 | 1 | 1
Intermittent claudication (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Ischaemia (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Microangiopathy (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 3 | 0 | 3 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 7 | 6 | 7 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 3 | 3 | 3 | 3 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 2 | 0 | 2 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 2 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Venous insufficiency (Vascular disorders) | 0 | 1 | 0 | 1 | 1
Venous thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Femoral artery embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Arteriosclerosis obliterans (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Colposcopy (Investigations) | 0 | 1 | 0 | 0 | 0
Endoscopy upper gastrointestinal tract (Investigations) | 0 | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoxic encephalopathy (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 1 | 4 | 1 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eplerenone: Double-blind Phase (May 25, 2010 Data Cut-off) (N=1360) | Placebo: Double-blind Phase(May 25, 2010 Data Cutoff) (N=1369) | Eplerenone: Double-blind Phase (N=1364) | Placebo: Double-blind Phase (N=1372) | Eplerenone: Open Label Phase (N=1245)
Atrial fibrillation (Cardiac disorders) | 29 | 36 | 37 | 42 | 42
Cardiac failure (Cardiac disorders) | 69 | 99 | 84 | 107 | 29
Constipation (Gastrointestinal disorders) | 27 | 13 | 30 | 15 | 0
Diarrhoea (Gastrointestinal disorders) | 30 | 40 | 35 | 46 | 0
Nausea (Gastrointestinal disorders) | 29 | 38 | 30 | 39 | 0
Chest pain (General disorders) | 33 | 29 | 35 | 33 | 0
Fatigue (General disorders) | 37 | 47 | 38 | 53 | 36
Oedema peripheral (General disorders) | 43 | 59 | 52 | 66 | 32
Bronchitis (Infections and infestations) | 47 | 44 | 54 | 52 | 0
Nasopharyngitis (Infections and infestations) | 45 | 41 | 49 | 48 | 28
Upper respiratory tract infection (Infections and infestations) | 35 | 31 | 28 | 34 | 25
Gout (Metabolism and nutrition disorders) | 26 | 31 | 30 | 36 | 28
Hyperkalaemia (Metabolism and nutrition disorders) | 95 | 43 | 101 | 48 | 38
Hypokalaemia (Metabolism and nutrition disorders) | 14 | 27 | 14 | 29 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 35 | 35 | 29 | 0
Dizziness (Nervous system disorders) | 53 | 56 | 64 | 62 | 43
Headache (Nervous system disorders) | 28 | 29 | 34 | 32 | 0
Renal impairment (Renal and urinary disorders) | 35 | 20 | 45 | 27 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 50 | 41 | 56 | 47 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 | 45 | 54 | 49 | 38
Pruritus (Skin and subcutaneous tissue disorders) | 29 | 15 | 29 | 15 | 0
Hypertension (Vascular disorders) | 23 | 36 | 28 | 37 | 0
Hypotension (Vascular disorders) | 43 | 31 | 53 | 33 | 33
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 28 | 26 | 0
insomnia (Psychiatric disorders) | 0 | 0 | 24 | 31 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 32
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 29 | 28 | 30
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 43
Urinary tract infection (Infections and infestations) | 0 | 0 | 28 | 26 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.